CLINICAL TRIAL: NCT05348681
Title: A Randomized, Double-blinded, Placebo-controlled, Phase 2a Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects With Hidradenitis Suppurativa
Brief Title: A Study to Evaluate RIST4721 in Hidradenitis Suppurativa (HS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to safety findings in ongoing Phase 2 trials.
Sponsor: Aristea Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIST4721-221
Record Dates: First submitted 2022-04-19; First posted 2022-04-27 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RIST4721 400 mg (Experimental): RIST4721 400 mg: 4 active (100 mg) tablets once daily for 12 weeks
  Interventions: Drug: RIST4721
- Placebo (Placebo Comparator): Placebo: 4 placebo tablets once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RIST4721 — RIST4721 tablets, 100 mg are blue, oval, biconvex film-coated tablets
  Arms: RIST4721 400 mg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-blinded, Placebo-controlled, Phase 2a Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects with Hidradenitis Suppurativa

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS for at least 1 year prior to screening
* HS lesions must be present in at least 2 distinct anatomic areas
* A total AN count (sum of abscesses and inflammatory nodules) > 6 across all anatomical sites at both the screening and baseline visits
* Willing to use contraception for the duration of the study

Exclusion Criteria:

* Presence of other skin conditions which may interfere with study assessments
* Presence of active, chronic or latent bacterial, viral, fungal mycobacterial infection (including latent TB) or history of infection within 4 weeks of screening
* Body Mass Index (BMI) >48kg/m2
* Breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Cahaba Dermatology & Skin Center, Birmingham, Alabama
  - Investigate MD, LLC, Scottsdale, Arizona
  - USC IDS Pharmacy, Los Angeles, California
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - ForCare Clinical Research, Tampa, Florida
  - The Indiana Clinical Trials Center, P.C., Plainfield, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wright State Physicians, Fairborn, Ohio
  - Progressive Clinical Research, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (2):
  - Enverus Medical Research, Surrey, British Columbia
  - SKiN Health, Cobourg, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RIST4721 400 mg | Placebo
Started | 17 | 8
Completed | 4 | 2
Not Completed | 13 | 6
Not completed — Study terminated by Sponsor | 8 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIST4721 400 mg | Placebo | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 8 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 14 | 5 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 1 | 4
  United States | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of TEAEs
Time Frame: Baseline to Week 12 (or end of study participation)
Population: Subjects with at least one TEAE
Measure: Count of Participants; unit: Participants
Arm/Group | RIST4721 400 mg | Placebo
Number analyzed (Participants) | 17 | 8
Participants | 9 | 4

2. Primary Outcome: Incidence of SAEs
Time Frame: Baseline to Week 12 (or end of study participation)
Population: Subjects with at least one SAE
Measure: Count of Participants; unit: Participants
Arm/Group | RIST4721 400 mg | Placebo
Number analyzed (Participants) | 17 | 8
Participants | 1 | 1

3. Secondary Outcome: Proportion of Subjects Achieving HiSCR50 at Week 12
Time Frame: Baseline to Week 12
Population: Subjects who completed Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | RIST4721 400 mg | Placebo
Number analyzed (Participants) | 7 | 3
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: From ICF signature to end of study participation.
Arm/Group | RIST4721 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/8
Other Adverse Events (participants affected / at risk) | 9/17 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIST4721 400 mg (N=17) | Placebo (N=8)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIST4721 400 mg (N=17) | Placebo (N=8)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT05348681/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05348681/SAP_001.pdf